CLINICAL TRIAL: NCT04803578
Title: The Effectiveness of Rehabilitation in Gait Recovery After Knee or Hip Arthroplasty: a Pilot Observational Study Based on Kinematic and Kinetic Parameters
Brief Title: The Effectiveness of Rehabilitation in Gait Recovery After Knee or Hip Arthroplasty
Acronym: Fast-Track2
Status: Completed | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Other Study IDs: JP-003
Record Dates: First submitted 2021-03-04; First posted 2021-03-17 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee
Keywords: Physical Therapy Modalities; Gait Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Knee Arthroplasty Group: Subjects that received knee arthroplasty 2-3 days before admission to undergo a rehabilitation period in our rehabilitation hospital.
  Interventions: Other: Conventional physiotherapy
- Hip Arthroplasty Group: Subjects that received hip arthroplasty 2-3 days before admission to undergo a rehabilitation period in our rehabilitation hospital.
  Interventions: Other: Conventional physiotherapy
- Age-Matched healthy Group: Subjects age-matched with those included in the knee and hip group. Subjects are asked to walk at their self-selected speed and at low speed matchable with those of the knee and hip group

INTERVENTIONS:
Other: Conventional physiotherapy — The subjects will receive rehabilitation according to the guidelines on the management of subjects after knee or hip arthroplasty, recovery of joint Range of Motion, recovery of lower limb strength, education to the crutches management, and stairs climbing and descending
  Groups: Hip Arthroplasty Group; Knee Arthroplasty Group

SUMMARY:
This study aims to evaluate the effectiveness of rehabilitation on gait recovery in subjects after knee or hip arthroplasty. Assessment is performed the day after admission (T0) and the day of discharge (T1), in a post-acute rehabilitation hospital, through an optoelectronic system (BTS DX-400). Other functional scales are administered to the subjects. during the rehabilitation period, subjects received conventional physiotherapy.

ELIGIBILITY:
Knee and Hip Arthroplasty subjects

Inclusion Criteria:

* Subjects > 18 years;
* Both Sexs;
* Knee or Hip Arthroplasty in the previous 3-4 days before admission;
* Subjects with clinical stability at admission (Hemoglobin > 9 g/l).

Exclusion Criteria:

* Fever at admission;
* Any rheumatic or systemic diseases;
* Previous surgery at the lower limbs (6 months before admission) or other arthroplasties at the lower limbs;
* MiniMental State Examination < 24;
* Other neurologic disorders.

For the healthy volunteers

Inclusion Criteria:

* Subjects age-matched with the subjects in the hip and knee group.

Exclusion Criteria:

* Any disorder that could negatively affect gait perfomance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this study, we included subjects who underwent in the previous 3/4 days for knee or hip arthroplasty subjects, before admission to our post-acute rehabilitation hospital, where they receive conventional physiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Gait Profile Score | From Admission (T0) up to 15/21 days (discharge) (T1)
  Change from Admission of Gait Profile Score untill 15/21 days (Discharge)
Change in Gai Deviation Index | From Admission (T0) up to 15/21 days (discharge) (T1)
  Change from Admission of Gait Deviation Index untill 15/21 days (Discharge)
Change in Gait Variable Scores | From Admission (T0) up to 15/21 days (discharge) (T1)
  Change from Admission of Gait Variable Score untill 15/21 days (Discharge)
Change in gait speed | From Admission (T0) up to 15/21 days (discharge) (T1)
  Change from Admission of Spatio-Temporal parameters untill 15/21 days (Discharge)
Change in gait cycle length | From Admission (T0) up to 15/21 days (discharge) (T1)
  Change from Admission of Spatio-Temporal parameters untill 15/21 days (Discharge)
Change in step length | From Admission (T0) up to 15/21 days (discharge) (T1)
  Change from Admission of Spatio-Temporal parameters untill 15/21 days (Discharge)
Change in gait cadence | From Admission (T0) up to 15/21 days (discharge) (T1)
  Change from Admission of Spatio-Temporal parameters untill 15/21 days (Discharge)
Change in gait cycle duration | From Admission (T0) up to 15/21 days (discharge) (T1)
  Change from Admission of Spatio-Temporal parameters untill 15/21 days (Discharge)
Change in stance phase duration | From Admission (T0) up to 15/21 days (discharge) (T1)
  Change from Admission of Spatio-Temporal parameters untill 15/21 days (Discharge)
Change in swing phase duration | From Admission (T0) up to 15/21 days (discharge) (T1)
  Change from Admission of Spatio-Temporal parameters untill 15/21 days (Discharge)
Change in single support phase duration | From Admission (T0) up to 15/21 days (discharge) (T1)
  Change from Admission of Spatio-Temporal parameters untill 15/21 days (Discharge)
Change in double support phase duration | From Admission (T0) up to 15/21 days (discharge) (T1)
  Change from Admission of Spatio-Temporal parameters untill 15/21 days (Discharge)

SECONDARY OUTCOMES:
Change in Modified Barthel Index | From Admission (T0) up to 15/21 days (discharge) (T1)
  Change from Admission of Modified Bathel Index untill 15/21 days (Discharge)
Change in International Knee Society score | From Admission (T0) up to 15/21 days (discharge) (T1)
  Change from Admission of International Knee Society score untill 15/21 days (Discharge)
Change in Merlè D'Aubigne score | From Admission (T0) up to 15/21 days (discharge) (T1)
  Change from Admission of Merlè D'Aubigne score untill 15/21 days (Discharge)
Change in Numerical Pain Rating Scale | From Admission (T0) up to 15/21 days (discharge) (T1)
  Change from Admission of Numerical Pain Rating Scale untill 15/21 days (Discharge)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pollet J, Pullara R, Bianchi LNC, Falso MV, Gobbo M, Buraschi R. Gait improvements in the early post-surgery rehabilitation phase in subjects receiving a total knee or hip arthroplasty: A prospective study. Gait Posture. 2025 Jul;120:25-33. doi: 10.1016/j.gaitpost.2025.03.024. Epub 2025 Mar 27. PMID 40179654